CLINICAL TRIAL: NCT06576635
Title: LUNG-05: Investigating Chemotherapy Effectiveness for NSCLC Metastatic Patients
Brief Title: LUNG-05: Investigating Chemotherapy Effectiveness for Non-Small Cell Lung Cancer (NSCLC) Metastatic Patients
Acronym: LUNG-05
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Frank Weinberg, Principal Investigator, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0301
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: NSCLC
MeSH Terms: interventions — Docetaxel; Paclitaxel; Gemcitabine; Pemetrexed; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Other): OncoChoiceTM results will provide ranking of drug effectiveness (e.g., active, inactive, moderately active drug) across a list of pre-selected chemotherapies (FDA-approved NSCLC treatments
  Interventions: Drug: Docetaxel; Drug: Paclitaxel; Drug: Gemcitabine; Drug: Pemetrexed; Drug: Vinorelbine

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m2 IV over 1-hour Day 1 of each 21-day cycle
Drug: Paclitaxel — 135 mg/m2 IV over 3 hours Day 1 of each 21-day cycle
Drug: Gemcitabine — 1000 mg/m2 IV over 30 minutes on Days 1, 8, and 15 of each 28-day cycle or 1,250 mg/m2 IV over 30 minutes on Days 1 and 8 of each 21 day cycle
Drug: Pemetrexed — 500 mg/m2 IV over 10 minutes on Day 1 of each 21-day cycle
Drug: Vinorelbine — 30 mg/m2 IV through a weekly injection over 6-19 minutes on Days 1, 8, and 15 of each 21-day cycle

SUMMARY:
This is a Single arm, Simon's two stage pilot study in which patients with Non-Small Cell Lung Cancer (NSCLC) with metastatic disease 2L and beyond will receive OncoChoice-informed chemotherapy following National Cancer Care Network (NCCN) treatment guidelines on dosage and scheduling for NSCLC FDA approved drugs.

DETAILED DESCRIPTION:
This is a Single arm, Simon's two stage pilot study in which patients with Non-Small Cell Lung Cancer (NSCLC) with metastatic disease 2L and beyond will receive OncoChoice-informed chemotherapy following National Cancer Care Network (NCCN) treatment guidelines on dosage and scheduling for NSCLC FDA-approved drugs. After confirmation of patient eligibility and patient consent receival, patients will undergo biopsy and/or removal of malignant fluids (paracentesis/ thoracentesis/ PleurX catheter) as part of standard of care procedures. Biosamples will be shared in a timely fashion (within 24 hr post collection) with study sponsors (OncoOptima) to test drug responsiveness. Participants will undergo additional testing as deemed necessary by the treating provider. Any additional treatments will be at the discretion of the treating provider.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age at time of consent
* ECOG performance status score of ≤2
* Advanced non-small cell lung cancer to meet histologically confirmed Stage IV NSCLC documented by biopsy.
* Patients have received at least 1 prior line of systemic therapy for Stage IV NSCLC, including but not limited to targeted therapy, and are currently candidates for 2L or later SOC chemotherapy. Exceptionally, patients with Stage III NSCLC who have received at least 1 line of systemic therapy may be considered eligible, pending principal investigator approval.
* Demonstrates adequate organ function; labs must be within treatment parameters for the individual institutional treatment plans for specific therapeutic agents. All screening labs to be obtained within 30 days prior to registration.
* Must have not received any cancer treatment for at least 2 weeks.
* Must be a candidate for small molecule drug treatment.
* Participants or their LAR must be able to provide written informed consent and HIPAA authorization for release of personal health information, via an approved UIC Institutional Review Board (IRB) informed consent form and HIPAA authorization.
* Women of childbearing potential must not be pregnant or breast-feeding. A negative serum or urine pregnancy test is required per institutional practice guidelines.
* As determined at the discretion of the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

* Active infection requiring systemic therapy within 7 days of enrollment.
* Uncontrolled HIV/AIDS or active viral hepatitis (e.g., HBV, HCV)
* Any ongoing significant toxicity resulting from prior anticancer therapy that, as determined by the treating provider, has the potential to interfere with the safety or efficacy assessment of this investigational regimen.
* ECOG performance status score >2
* Clinically significant lung, heart, or autoimmune disease
* Life expectancy <12 weeks
* Prior solid organ or bone marrow transplant
* Antibiotics, live vaccines or other type of surgery within 4 weeks prior intervention treatment
* Pregnant or nursing
* Any prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of this investigational regimen, as determined by the treating provider.
* Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial.
* Another major comorbidity, as determined by treating provider.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
To estimate the objective response rate (ORR) as measured by investigator assessment in patients with metastatic NSCLC treated with at least 2L of chemotherapy who have had OncoChoice-informed treatment | Every 6-8 weeks through study completion, an average of 2 years
  The objective response rate is the proportion of all subjects with confirmed PR or CR according to investigator assessment, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment).

SECONDARY OUTCOMES:
To estimate the 6-month progression-free survival (PFS) in 2L and beyond NSCLC patients who receive OncoChoice-informed chemotherapy regimen | Day 1 of treatment through study completion, an average of 2 years
  PFS is defined as the time from D1 of treatment until the criteria for disease progression is met as defined by investigator-assessed criteria or death as a result of any cause.
To estimate the overall survival (OS) in 2L and beyond NSCLC patients who receive OncoChoice-informed chemotherapy regimen | Day 1 of treatment through study completion, an average of 2 years
  OS is defined as the time from D1 of treatment to death as a result of any cause.
To describe changes in health-related quality of life (HRQoL) over the course of treatment following OncoChoice-informed regimen vs. standard chemotherapy | Screening through study completion, an average of 2 years
  Changes in health-related quality of life (HRQoL) will be studied using self-reported and validated questionnaires that address addressing physical, physiological, emotional, and social issues

OTHER OUTCOMES:
To characterize changes in blood circulating immune cell populations before and after OncoChoice-based treatment by utilizing spectral flow analysis | Day 1 of treatment through study completion, an average of 2 years
  Circulating blood immune cell populations will be determined by spectral flow analysis
To explore blood circulating cytokine levels before and after OncoChoice based treatment by utilizing bulk cytokine analysis (Bruker Cellular Analysis). | Day 1 of treatment through study completion, an average of 2 years
  Circulating blood cytokine levels determined utilizing bulk cytokine analysis (Bruker Cellular Analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Weinberg, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Cancer Center, Chicago, Illinois, United States